CLINICAL TRIAL: NCT00737191
Title: Analgesic Effect of Olanzapine in Cancer Pain: A Double-Blind Randomized Placebo-Controlled Parallel Group Pilot Study
Brief Title: Opioids With or Without Olanzapine in Treating Patients With Moderate to Severe Cancer Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No accrual; No patients enrolled
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Eric E. Prommer, M.D., Mayo Clinic Cancer Center
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000588630; P30CA015083 (NIH); MCS930 (Other: Mayo Clinic Cancer Center); 07-007571 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Hematopoietic/Lymphoid Cancer; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; hematopoietic/lymphoid cancer; pain
MeSH Terms: conditions — Hematologic Neoplasms; Pain | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Active Comparator): Patients receive oral opioid and oral placebo once daily for 4 weeks.
  Interventions: Other: placebo
- Arm II (Experimental): Patients receive oral opioid and 2.5 mg oral olanzapine once daily for 4 weeks.
  Interventions: Drug: olanzapine
- Arm III (Experimental): Patients receive oral opioid and 5 mg oral olanzapine once daily for 4 weeks.
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: olanzapine — Given orally
  Arms: Arm II; Arm III
Other: placebo — Given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Opioids lessen pain caused by cancer. It is not yet known whether opioids are more effective when given together with or without olanzapine in treating cancer pain.

PURPOSE: This randomized clinical trial is studying opioids to see how well they work when given together with or without olanzapine in treating patients with moderate to severe cancer pain.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the analgesic effect of olanzapine when administered in combination with opioids in patients with cancer pain.
* To assess the opiod-sparing effect of olanzapine vs placebo.
* To assess the effect of olanzapine on opioid adverse effects.

OUTLINE: Patients undergo opioid titration with a step 3 opioid to maintain a less than 4/10 level of pain (on a 0-10 numeric pain rating scale) to establish a opioid starting dose. When the pain rating increases, patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive oral opioid and oral placebo once daily for 4 weeks.
* Arm II: Patients receive oral opioid and 2.5 mg oral olanzapine once daily for 4 weeks.
* Arm III: Patients receive oral opioid and 5 mg oral olanzapine once daily for 4 weeks.

Patients undergo quality of life assessments at baseline and three times weekly by questionnaires using a scale from 0-3 and pain assessments periodically by Brief Pain Inventory, Edmonton Symptom Assessment Scale, Linear Analogue Scale Assessments, and Mini-Mental State Examination.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Moderate to severe cancer pain

  * Pain score ≥ 7/10 (0-10 numeric pain rating scale)
  * Requires strong opioids (step 3) for pain control or are already on stable doses of step 3 opioids
* Opioid induced cognitive dysfunction or cognitive impairment, defined as cognitive disorder not otherwise specified according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) allowed
* No nonmalignant pain

  * If patient has both malignant and nonmalignant pain, eligibility will be determined by the predominant site of pain

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 3 months
* Normal renal function
* Not pregnant or nursing
* Negative pregnancy test
* Must have a telephone
* Able to complete patient questionnaires alone or with assistance
* No delirium
* No hepatic dysfunction
* No nursing home patients
* No intractable nausea or vomiting
* No true allergy or intolerance to opioids
* No gastrointestinal pathology that influences absorption of opioids
* No drug seeking behavior or recent substance abuse history
* No major depression
* No respiratory compromise
* No evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* No evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study

PRIOR CONCURRENT THERAPY:

* More than 1 month since prior radiotherapy, chemotherapy, or radionuclides
* More than 1 month since prior bisphosphonates
* No prior surgery that influences absorption of opioids
* No concurrent therapeutic procedures or treatments that influence pain
* No concurrent active radiation or antineoplastic therapies
* No concurrent retroviral therapies
* No concurrent drugs that interfere with CYP34A, CYP1A2, or CYP2D6
* No concurrent drugs that interfere with morphine metabolism
* No concurrent medications that will influence the disposition of morphine or methadone
* No other concurrent antiemetics, antianxiety, or neuroleptic agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Two-point pain improvement from baseline (0-10 numeric pain rating scale)

SECONDARY OUTCOMES:
Comparison of active treatment vs placebo
Effect of olanzapine on opiod adverse effects
Relationships between endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Eric E. Prommer, MD, Study Chair — Mayo Clinic